CLINICAL TRIAL: NCT06718114
Title: A Study on Early Removal of Urinary Catheter After Gastric Cancer Surgery Applying ERAS Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nanjing University of Chinese Medicine (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021NL-167-02; JD201807 (Other Grant/Funding Number: China Medical Education Association)
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Urinary Catheter Removal After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate removal of urinary catheter (Experimental): The urinary catheter will be removed immediately after surgery.
  Interventions: Procedure: immediate urinary catheter removal
- early removal of urinary catheter (Other): The urinary catheter will be kept after surgery and be removed within 48 hours after surgery.
  Interventions: Procedure: early removal of urinary catheter

INTERVENTIONS:
Procedure: immediate urinary catheter removal — Immediate urinary catheter removal indicates that the urinary catheter will be removed immediately after surgery.
  Arms: immediate removal of urinary catheter
Procedure: early removal of urinary catheter — The urinary catheter will be kept after surgery and be removed within 48 hours after surgery.
  Arms: early removal of urinary catheter

SUMMARY:
This study compared the immediate removal of urinary catheter and early removal of urinary catheter after radical gastrectomy to explore the feasibility of immediate removal of urinary catheter after radical gastrectomy, especially in the incidence of urinary retention, whether immediate removal is not inferior to early removal.

ELIGIBILITY:
Inclusion Criteria:

* underwent elective radical gastrectomy
* applied ERAS protocols during perioperative period
* aged 18～80 years old

Exclusion Criteria:

* benign prostatic hyperplasia
* urinary system stones, tumors, strictures, deformities or surgeries
* pelvic surgery history
* abnormal preoperative urine routine
* medication intake that affects urination function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative urinary retention incidence | From urinary catheter removed to 6 hours after removal

SECONDARY OUTCOMES:
postoperative urinary tract infection incidence | from postoperative day 1 to postoperative day 7
anxious status | postoperative day 1
  measured by Kolcaba scale, Kolcaba scale scores from 30 to 112, higher scores mean the patients feel more comfortable during hospitalization (a better outcome).
comfort status | postoperative day 1
  measured by hospital anxiety and depression scale (HAD scale), HAD scale scores from 0 to 20, a higher score means the patients feel more stressful during hospitalization (a worse result).

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei C, Wang G, Wang HF, Pan HF, Jiang ZW, Qu MW. Immediate versus early urinary catheter removal after gastrectomy under enhanced recovery after surgery protocols: randomized clinical trial. BJS Open. 2025 Jul 1;9(4):zraf088. doi: 10.1093/bjsopen/zraf088. PMID 40827509